CLINICAL TRIAL: NCT03044769
Title: Follow up of Congenital Lung Anomalies (CLA) With Antenatal Diagnosis - a Swiss Multicentric Database
Brief Title: Congenital Lung Anomalies (CLA) Swiss Database
Acronym: CLADatabase
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Isabelle Ruchonnet-Métrailler, Principal Investigator, University Hospital, Geneva
Other Study IDs: CLA-2016
Record Dates: First submitted 2017-01-31; First posted 2017-02-07 (Estimated); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Congenital Lung Malformation; Congenital Lung Cyst; Sequestrum; Bronchogenic Cancer; Pleuropulmonary Blastoma; Acinar Dysplasia
Keywords: Congenital Lung Anomalies
MeSH Terms: conditions — Cystic Adenomatoid Malformation of Lung, Congenital; Pleuropulmonary blastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — To create a biobank with the different samples of patients undergoing surgery, healthy edge of resections being considered as control tissue. Leukocyte DNA will be compared with lung tissue DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with CLA with surgery
  Interventions: Procedure: Malformations resection
- Patient with CLA without surgery

INTERVENTIONS:
Procedure: Malformations resection — Resection of the malformation lung sections with a healthy adjacent part
  Groups: Patient with CLA with surgery

SUMMARY:
Congenital lung anomalies include different pathologies such as congenital cystic adenomatoid malformation, pulmonary sequestration, bronchial atresia, emphysema, bronchogenic cyst. They concern less than 1/10000 births and their physiopathological origin is still poorly understood. The main goal of this project is to pool the cases from different swiss centers on a prospective cohort study, first to increase knowledge of clinical and radiological evolution and their correlation with histological data, and second to analyse the pathological embryological mechanism underlying these malformations.

DETAILED DESCRIPTION:
1. To register prospectively clinical, biological, radiological and histological datas in a multicentric database (secured internet link, via Secutrial® software). for children with prenatal diagnosis of this kind of malformation. This study is conducted by a multidisciplinary team, involving obstetricians, neonatologists, pneumologists, pediatric surgeons, radiologists and anatomopathologists.
2. To create a tissue biobank

Outcomes:

1. Contribute to the definition of a standardized procedure at the Swiss level for the treatment of patients suffering from these malformations,
2. Improve the assessment of lesion evolution related to CLA, and
3. Possibly validate some biomarkers, which could help to identify individuals at risk. On the long term, these results could also support the development of innovative therapies targeting the factors involved in lung development.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with congenital lung anomalies

Exclusion Criteria:

* None

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Recruitment for this study is performed through a discussion with parents of the child during prenatal and postnatal medical consultations.
  Blood samples will be collected during surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in clinical of patients with CLA between different time point | Birth, 1 month of life, 4 months of life, 9-18 months of life, 6 months post surgery, 1 year post surgery, 7 years old, 10 years old, 12 years old
  Clinical measurements: size (cm), weight (kg), saturation (%)
Analysis of CLA physiopathology | samples collected during surgery
  Analysis of growth factors, transcription factors and extracellular components implicated in CLA genesis by immunohistochemistry, transcriptomic and proteomic methods
Change in lung function | 7 years old,10 years old, 12 years old, 16 years old
  FEV1 (l/min), FEV1/FVC (%)TLC (L) DLCO (ml/min/mmHg)
Change in Scar aspect and thoracic deformation of patients with CLA between different time point | 6 months post surgery, 1 year post surgery, 7 years old, 10 years old, 12 years old
  Description
Change in lung radiological images of patients with CLA between different time point | 1 month of life, 4 months of life, 9-18 months of life, 6 months post surgery, 1 year post surgery, 7 years old, 10 years old, 12 years old
  Chest X-ray and Thoracic CT Scan lesion description
Change in lesion size described by antenatal ultrasound of patients with CLA between different time point | 22, 28, 32 and 37 weeks of gestation
  lesion size (mm) CVR, estimated wight (gr), Head circumferences (cm)
Change in lesion description by antenatal ultrasound of patients with CLA between different time point | 22, 28, 32 and 37 weeks of gestation
  Lesion description (micro cysts, macrocysts),lesion localisation

SECONDARY OUTCOMES:
Report biomarkers implicated in CLA with a potential role in lesion oncogenic transformation | 1 year post surgery
  Comparison using exome analysis : CLA lesion, healthy adjacent part and blood DNA

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Andrieu Vidal, MD PhD, Principal Investigator — University Hospital, Geneva; Isabelle Ruchonnet-Métrailler, MD PhD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided